CLINICAL TRIAL: NCT07061431
Title: In Vitro and in Vivo Evaluation of the Anti-Inflammatory and Antithrombotic Efficacy of Natural Bioactives in Human Platelets
Brief Title: In Vitro and in Vivo Evaluation of the Anti-Inflammatory and Antithrombotic Synergy of Vitamin C and Bioflavonoids in Healthy Subjects
Acronym: VCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Alexandros Tsoupras, Assistant Professor, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ΔΠΘ/ΕHΔΕ/7690/70, 27-9-2024
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cardio-protection
Keywords: Anti-platelet; Anti-inflammatory; PAF; Thrombin; ADP; cardio-protective; platelet aggregation
MeSH Terms: interventions — Ascorbic Acid; Flavonoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VCF Group (Active Comparator): Group of healthy subjects that recieved orally a high dose (1 g) vitamin C supplement containing also a low dose (50 mg) citrus and rose bioflavonoids (VCF), for 28 days
  Interventions: Dietary Supplement: High Dose of Vitamin C with ir without 50 mg of flavonoids
- VC (Active Comparator): Group of healthy subjects that recieved orally a high dose (1 g) vitamin C supplement, for 28 days
  Interventions: Dietary Supplement: High Dose of Vitamin C with ir without 50 mg of flavonoids

INTERVENTIONS:
Dietary Supplement: High Dose of Vitamin C with ir without 50 mg of flavonoids — The anti-inflammatory and anti-platelet efficacy and synergy of a supplement containing high dose (1 g) of vitamin C and a low dose (50 mg) citrus and rose bioflavonoids (VCF), was assessed in platelets of blood samples collected from healthy subjects, prior the oral administration (t=0 days) and just after this administration for 1 month (VCF Group), VERSUS the findings from the same procedure contacted for a supplement containing only high dose (1 g) of vitamin C (VC Group)

SUMMARY:
This study aimed to evaluate the antioxidant potential, and especially the anti-inflammatory and antiplatelet biological efficacy and synergy of a high dose (1 g) vitamin C - low dose (50 mg) bioflavonoid (VCF) based supplement using both in vitro approaches and an and in vivo clinical trial in human platelets from healthy subjects administered orally for 1 month the VCF supplement (VCF Group) versus the administration of a 1 g vitamin C supplement (VC Group).

DETAILED DESCRIPTION:
For the In vivo clinical study, blood samples were collected from all participants at baseline (day 0), prior to supplementation (t = 0), and again after 28 days of daily supplementation of VC or VCF. Platelet aggregation was evaluated using three agonists: platelet activating factor (PAF), ADP, and thrombin. Immediately after collection, blood samples collected in citrate containing monovette tubes were centrifuged at 194 × g for 18 minutes at 24 °C to isolate platelet-rich plasma (PRP). The remaining blood was subsequently centrifuged at 1465 × g for 20 minutes at 24 °C to obtain platelet-poor plasma (PPP). PRP and PPP were separated into distinct tubes for further analysis. For aggregometry assays, 250 μL of PRP containing a magnetic stir bar and 500 μL of PPP without stir bar were transferred to each aggregometer cuvette and placed at the appropriate positions at the aggregometer. Platelet aggregation was quantified by determining the mean EC₅₀ values, representing the concentration of each agonist required to induce 50% platelet aggregation. These values were normalized per gram of total content , vitamin C , and flavonoid content as regarding vitamin C and flavonoid supplement. The change in EC₅₀ values after 28 days of supplementation provided an indication of the supplement's modulatory effect on platelet aggregation

ELIGIBILITY:
Inclusion Criteria:

Subjects should:

* not have a pathological condition related to platelet and leukocyte activity
* not have a chronic pathological condition
* have a normal BMI
* not take medications that have anti-inflammatory and/or antithrombotic effects

Exclusion Criteria:

If Subjects

* have a pathological condition related to platelet and leukocyte activity
* have a chronic pathological condition
* not have a normal BMI
* take medications that have anti-inflammatory and/or antithrombotic effects

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Anti-platelet cardio-protective efficacy | 1 month
  The increase of the EC50 values of PAF/ADP/Thrombin induced platelet aggregation in the VCF Group versus the VC Group

CONTACTS AND LOCATIONS:
Locations (1):
- School of Chemistry, Faculty of Sciences, Democritus University of Thrace, Kavala, Kavala, Greece